CLINICAL TRIAL: NCT06448338
Title: MyDiaMate for Remission of Elevated Diabetes Distress in Type 1 Diabetes: the UK MyREMEDY Randomized Controlled Trial
Brief Title: UK MyREMEDY Clinical Trial
Acronym: UK-MyREMEDY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Forschungsinstitut der Diabetes Akademie Mergentheim (Other); University of Malaga (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 329634; RMS360 (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyDiaMate (Experimental): 2/3 of participants will be randomized into this arm. They will receive access to MyDiaMate for 6 months.
  Interventions: Behavioral: MyDiaMate
- Care as Usual (No Intervention): 1/3 of participants will be randomized into this arm. They will continue their care as usual for 3 months. After 3 months, they receive access to MyDiaMate if desired.

INTERVENTIONS:
Behavioral: MyDiaMate — MyDiaMate program
  Arms: MyDiaMate

SUMMARY:
The UK MyREMEDY study investigates whether MyDiaMate, an online self-help program, can effectively improve the mental health of adults with type 1 diabetes compared to those receiving care as usual.

DETAILED DESCRIPTION:
The psychological burden of living with and self-managing type 1 diabetes is well-recognized. Nevertheless, access to mental health services for people with type 1 diabetes is generally limited, even in well-resourced settings. Digital solutions or e-mental health, a rapidly expanding field, offer a complement to existing services. However, while many apps target glucose and lifestyle, particularly for type 2 diabetes, few digital tools focusing on healthy coping and mental health for type 1 diabetes exist. MyDiaMate was developed to alleviate this deficiency and its effectiveness (in terms of reduction of diabetes distress among people with type 1 diabetes) will be evaluated by this study. UK MyREMEDY is conducted in conjunction with a wider evaluation of MyDiaMate in the Netherlands, Spain, and Germany.

Previously, an observational pilot study in the Netherlands demonstrated the acceptability and feasibility of MyDiaMate and additionally suggested positive effects on mental health. Nevertheless, MyDiaMate has not been evaluated in a UK setting. The principal research objective of this study is to determine the effectiveness of MyDiaMate over time in adults with type 1 diabetes. This will be assessed in terms of improvement of mental health, with diabetes distress as primary outcome, relative to care as usual.

The effectiveness of MyDiaMate will be tested in a two-arm parallel randomized controlled trial. This study design will allow researchers to assess differences in mental health, diabetes self-care, and glycemic control in participants using MyDiaMate versus participants undergoing care as usual (randomized 2:1).

The study population will consist of adults with type 1 diabetes in the UK who were diagnosed at least 6 months prior and who experience distress related to their diabetes. After participants are screened for eligibility and confirm their participation in the study, they will complete a baseline assessment and be randomized to the intervention or control group. For their first 3 months of participation, the control group will receive care as usual, while the participants in the experimental group will be given access to MyDiaMate via an online link. After 3 months, all participants irrespective of randomized groups will be given access to MyDiaMate. Access to MyDiaMate will end after 6 months of study participation. All participants will additionally be asked to complete several online, self-reported measures of primary and secondary outcomes at baseline, three months, and six months.

MyDiaMate offers online modules centered around common sources of diabetes distress, such as the disruptive impact of stress on blood glucose, fear of hypoglycemia, worries about complications, disordered eating, and stressful social interactions, as well as low wellbeing and fatigue. Grounded in principles of cognitive behavioral therapy, MyDiaMate includes psycho-education and coping strategies, presented in a variety of formats, including written content, videos, diaries, and other activities. The participants can access the program on their personal device as often as wished for the duration of the study with no prescribed frequency of use.

Participation in this study is low risk and participants have the opportunity to engage with MyDiaMate as much as desired. Completion of the study questionnaires is estimated to take 2 hours, spread across the participation period (6 months). The participants may benefit from use of MyDiaMate and experience improved mental health and reduced diabetes distress.

After the study has concluded in the UK, the investigators will share the anonymized data with the research team of the international MyREMEDY clinical trial. Subsequent pooled analyses will contribute to complete evaluation of MyDiaMate and the further support of the mental wellbeing of people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at signing the informed consent form
* Type 1 diabetes diagnosis at least 6 months ago
* Having access to the internet and a smartphone/tablet/laptop/computer for the entirety of study participation
* Experiencing diabetes distress (checked during a phone call between research assistant and participant. The condition is met if the participant has an average score of ≥2 on the 2-item Diabetes Distress Scale [DDS-2], representing clinically meaningful diabetes distress)

Exclusion Criteria:

* Having been diagnosed with a psychiatric disorder in the past 6 months for which the person is under psychological/psychiatric treatment
* Suicidality
* Having started a treatment with psychotropic medication in the past 3 months
* Cannot read and speak English
* Experience of cognitive problems that hamper using MyDiaMate or vision/auditory problems that are hindering in daily life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Diabetes Distress will be assessed at 0 months (baseline), 3 months (intervention effects), and after 6 months (follow-up).
  Diabetes Distress will be assessed through the 20-item Problem Areas In Diabetes questionnaire (PAID-20). The PAID questionnaire measures diabetes distress on a 5-point Likert scale ranging from 1 (not a problem) to 5 (serious problem). A higher score represents higher diabetes distress.

SECONDARY OUTCOMES:
Emotional well-being | Emotional well-being will be assessed at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Emotional well-being will be operationalised as the score on the 5-item World Health Organization Well-Being Index (WHO-5). The score on the WHO-5 is measured on a 6-point scale ranging from 0 (at no time) to 5 (all of the time), with a lower score representing less emotional well-being.
Psychological self-efficacy in relation to diabetes | Psychological self-efficacy in relation to diabetes will be assessed at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Operationalised through the short form of the Diabetes Empowerment Scale (DES-SF). Psychological self-efficacy in relation to diabetes is assessed on a 5-point scale ranging from 0 (strongly disagree) to 4 (strongly agree), with higher scores representing higher psychological self-efficacy in relation to diabetes.
Social engagement | Social engagement will be measured at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Social engagement will be assessed through the 6-item Lubben Social Network Scale (LSNS-6). The LSNS measures social engagement on a 6-point scale ranging from 0 (none) to 5 (nine or more). A higher score represents higher social engagement.
Fatigue | Fatigue will be measured at 0 months (baseline), 3 months (intervention effects), and 6 months (follow-up).
  Fatigue will be assessed through the 8-item Fatigue subscale of the Checklist Individual Strength (CIS-F). The CIS-F consists of both positively and negatively framed items that are measured on a 7-point scale ranging from 1 (no, that is not true) to 7 (yes, that is true). The positively framed items (e.g., I feel fit) will be reverse coded. A higher score will therefore represent stronger fatigue.
HbA1c | HbA1c will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up).
  Participants will self-report various outcome measures typical for assessing glycemic control in type 1 diabetes. One of these measures is the self-reported glycated hemoglobin (HbA1c) value. A lower score represents better glycemic control. For data analysis, all scores measured in percentage will be transformed to a HbA1c value measured in mmol/mol.
Time in/above/below range | Time in/above/below range will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up).
  Participants will self-report various outcome measures typical for assessing glycemic control in type 1 diabetes. One of these measures is the self-reported time in/above/below range. Participants can indicate their own personal target range for blood glucose values, and then indicate the percentage of time during which they were in, above, and below this personal range across the past 14 days. A higher percentage for time in range represents better glycemic control. A lower percentage for time above range and time below range represents worse glycemic control.
Events of ketoacidosis | Frequency of events of ketoacidosis will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up).
  Participants will self-report various outcome measures typical for assessing glycemic control in type 1 diabetes. One of these measures is the self-reported frequency of events of ketoacidosis in the past 12 months when measured at baseline, and in the past 3 months when measured at the 3 and 6 months assessment, respectively. A higher self-reported frequency of events of ketoacidosis represents worse glycemic control.
Events of severe hypoglycemia | Frequency of events of severe hypoglycemia will be self-reported at 0 months (baseline), 3 months (intervention effect), and 6 months (follow-up).
  Participants will self-report various outcome measures typical for assessing glycemic control in type 1 diabetes. One of these measures is the self-reported frequency of events of severe hypoglycemia in the past 12 months when measured at baseline, and in the past 3 months when measured at the 3 and 6 months assessment, respectively. A higher self-reported frequency of events of severe hypoglycemia represents worse glycemic control.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- See also: Link to study website — https://www.kcl.ac.uk/research/myremedytrial